CLINICAL TRIAL: NCT02535689
Title: Safety of Tofacitinib, an Oral Janus Kinase Inhibitor, in Systemic Lupus Erythematosus; a Phase Ib Clinical Trial and Associated Mechanistic Studies
Brief Title: Safety of Tofacitinib, an Oral Janus Kinase Inhibitor, in Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 150185; 15-AR-0185
Record Dates: First submitted 2015-08-28; First posted 2015-08-31 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-04-25

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Anti-DNA Antibody; Tofacitinib; Lupus; Safety
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Active Comparator): ARM 1: 10 of SLE patients will be heterozygous or homozygous for the STAT 4 risk alleles, receive treatment with tofacitinib 5 mg twice daily.
  Interventions: Drug: Tofacitinib
- 2 (Active Comparator): ARM 2: 10 of SLE patients will NOT be heterozygous or homozygous for the STAT 4 risk alleles, receive treatment with tofacitinib 5 mg twice daily.
  Interventions: Drug: Tofacitinib
- 3 (Placebo Comparator): ARM 3: 10 of SLE patients will be with variable genotypes will receive placebo twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tofacitinib — Oral administration of tofacitinib, 5 mg
  Arms: 1; 2
Drug: Placebo
  Arms: 3

SUMMARY:
Background:

Systemic lupus erythematosus (lupus) is an autoimmune disease that often involves many systems and organs of the body. Symptoms can include fever, joint pains, and rashes. Serious lupus can also damage organs like the kidneys, lungs, or brain. Drugs used for lupus can have serious side effects. Also, the drugs don t help some people. Researchers want to find new, more effective and safe treatments.

Objective:

To evaluate the safety and tolerability of the drug tofacitinib (study drug) in people with lupus.

Eligibility:

People ages 18 and older who have mild to moderate lupus and are not currently or haven t recently had certain lupus treatments.

Design:

Participants will be screened in another protocol.

Participants will have 7 five-hour visits over about 3 months. They will fill out multiple questionnaires. They will have tests, including:

* Physical exam
* Blood and urine tests
* ECG/EKG: Soft electrodes are stuck to the skin to monitor the heart.
* Optional SphygmoCor: Cuffs are attached to the arm and thigh to measure blood pressure and flow speed.
* Optional Endopat: A thimble-shaped cup is placed on the finger to measure blood flow. A cuff is put on the arm to measure blood pressure and flow.
* Optional CAVI: ECG electrodes are placed on both wrists, a microphone placed on the chest, and a blood pressure cuff placed on each arm and leg to measure blood pressure and velocity.

Participants will receive either the study drug or a placebo. They will take this twice a day by mouth for 56 days.

Participants will be contacted by phone 4 times....

DETAILED DESCRIPTION:
BACKGROUND:

Systemic Lupus Erythematosus (SLE) is an autoimmune disease with variegated clinical presentation resulting from involvement of multiple biologic pathways. The pathways that lead to loss of tolerance in SLE include: multiple autoreactive cell types (B, T, dendritic, Th17 and regulatory T cells) and abnormal cytokine milieus, genetic factors, environmental and hormonal influences, all of which can influence cell differentiation patterns and reset tolerance checkpoints. In addition, recent studies indicate a putative role for neutrophils in lupus pathogenesis and associated end-organ damage. Currently available therapeutics are frequently inadequate to treat disease flares and simultaneously expose patients to potentially serious toxicities. Further, premature cardiovascular disease not explained by the Framingham risk equation has become one of the most important causes of morbidity and mortality in this patient population. To date, no treatment used in lupus appears to significantly decrease cardiovascular risk. Identifying a drug that has immunomodulatory effects and is also vasculoprotective is an unmet need in this disease.

Tofacitinib is an orally administered Janus kinase (JAK) inhibitor that has recently been approved by the Food and Drug Administration for the treatment of moderate to severe rheumatoid arthritis (RA).

The JAKs are a family of intracellular enzymes (JAK1, 2 and 3 and TYK2) that mediate signaling via a broad range of cytokine receptors. Targeting JAKs is an attractive therapeutic possibility for SLE for many reasons. Many of the inflammatory cytokines implicated in the pathogenesis of SLE signal via the JAK-STAT pathways. JAK inhibitors have been found to have efficacy in various murine models of lupus. Mice treated with a JAK2 inhibitor exhibited reduced serum levels of IL-6, and IL-17 along with reduced numbers of long-lived autoantibody producing plasma cells in the spleen and bone marrow. Furthermore, we have found that administration of tofacitinib reduced serum levels of ANA, IL-6, and IFN-gamma; and ameliorated glomerulonephritis (unpublished data).

This study therefore represents an innovative investigative measure of the safety and efficacy of JAK inhibition in SLE that is predicted by genetic predisposition. We will also investigate effects of tofacitinib on vascular function in SLE subjects and identify biomarkers that may be useful as endpoints in future studies.

PRIMARY OBJECTIVE:

To determine the safety and tolerability of tofacitinib in patients with SLE and mild to moderate disease activity.

STUDY DESIGN:

This is a Phase Ib, randomized, double blind, placebo controlled clinical trial of orally administered tofacitinib, 5 mg twice daily, for the treatment of SLE subjects with mild to moderate disease activity stratified by the presence or absence of STAT4 risk alleles.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subject is capable of providing written informed consent.
* Subject is greater than or equal to 18 years old.
* Meets at least 4 of 11 modified American College of Rheumatology (ACR) (1997) Revised Criteria for the Classification of Systemic Lupus Erythematosus.
* Has mild to moderate disease activity defined as a SLEDAI 2K more than or equal to 2 and less than or equal to 14 at the screening visit.
* If on glucocorticoids, the dose must be less than or equal to 20 mg daily and stable for the 4 weeks prior to screening visit.
* If on hydroxychloroquine or other antimalarials such as chloroquine or quinacrine, the dose must have been stable for the 12 weeks prior to screening visit. The maximum allowed dose is hydroxychloroquine up to 400 mg/day or 6.5 mg/kg/day if more than 400 mg/day. The maximum allowed dose for chloroquine phosphate is up to 500 mg daily and for quinacrine up to100 mg daily.
* Males and females with potential for reproduction must agree to practice effective birth control measures. Females should be on adequate contraception if they are of child-bearing potential documented by a clinician, unless patients or spouse have previously undergone a sterilization procedure. Adequate will be considered intrauterine device (IUD) alone or hormone implants, hormone patches, injectables, or oral contraceptives plus a barrier method (male condom, female condom or diaphragm), abstinence or a vasectomized partner
* If patients are on ACE inhibitors or ARB medications, dose of this medication must be stable for 4 weeks prior to study entry.
* Patients may be on lipid lowering medications if initiated at least 6 months prior to the screening visit.

EXCLUSION CRITERIA:

* Pregnant or lactating women. Women of childbearing potential are required to have a negative pregnancy test at screening.
* Current or prior treatment with rituximab, belimumab or any other biologic agent in the 6 months prior to screening.
* Current treatment with immunosuppressive drugs (methotrexate, azathioprine, mycophenolate mofetil, cyclosporine, tacrolimus). Glucocorticoids are allowed as per the inclusion criteria. At the investigator s discretion, glucocorticoids may be tapered during the study.
* Patients previously on methotrexate, mycophenolate mofetil, cyclosporine or tacrolimus should have stopped it for at least 8 weeks at the time of screening.
* Treatment with cyclophosphamide, pulse methylprednisolone or IVIG within the 6 months prior to screening.
* Increase in glucocorticoid dose within 4 weeks of screening.
* A history of drug or alcohol abuse within the 6 months prior to screening.
* History of chronic liver disease or elevated LFTs:

  * ALT or AST greater than or equal to 2x upper limit of normal at screening
  * serum unconjugated bilirubin > 2mg/dL at screening
* Dialysis or serum creatinine >1.5mg/dL.
* Protein to creatinine ratio of more than 1 mg/mg or 24 hours urine protein of more than 1000 mg.
* Active urinary sediment (WBC, RBC or mixed cellular casts 1+ or more /hpf).
* Hypercholesterolemia: Values after an 8-12 hour fasting blood specimen: total cholesterol >250 mg/dL or LDL >180 mg/dl or hypertriglyceridemia (triglyceride >300 mg/dL) within plus or minus 45 days of screening visit.
* Active infection that requires the use of oral or intravenous antibiotics and has not resolved at least 2 weeks prior to the administration of the first dose of study medication.
* Active chronic infections including but not limited to HIV, Hepatitis B, Hepatitis C, and BK viremia at screening visit.
* History of cancer.
* Known active tuberculosis or untreated latent tuberculosis.
* History of opportunistic infections.
* Subjects with active renal or central nervous system disease or a BILAG A in any organ system.
* WBC <2500/Microlitre or ANC <1,000/Microlitre, Hgb <9.0 g/dL or platelets <70,000/Microlitre or absolute lymphocyte count < 500/Microlitre.
* Current treatment with potent inhibitors of Cytochrome P450 3A4 (CYP3A4) (e.g., ketoconazole) or receiving one or more concomitant medications that result in both moderate inhibition of CYP3A4 and potent inhibition of CYP2C19 (e.g., fluconazole) that would increase serum availability of tofacitinib. Past treatment with the above mentioned agent is allowed if it was more than a week prior to the administration of the first dose of study medication.
* Significant impairment of major organ function (lung, heart, liver, kidney) or any condition that, in the opinion of the Investigator, would jeopardize the subject s safety following exposure to the study drug.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-08-28; Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is safety of tofacitinib in SLE subjects. | 5 years

SECONDARY OUTCOMES:
Assessments of clinical response. | 5 years
  Assessment of biologic effects.
Assessment of biologic effects. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sarfaraz A Hasni, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] O'Shea JJ, Holland SM, Staudt LM. JAKs and STATs in immunity, immunodeficiency, and cancer. N Engl J Med. 2013 Jan 10;368(2):161-70. doi: 10.1056/NEJMra1202117. No abstract available. PMID 23301733
- [Background] O'Shea JJ, Laurence A, McInnes IB. Back to the future: oral targeted therapy for RA and other autoimmune diseases. Nat Rev Rheumatol. 2013 Mar;9(3):173-82. doi: 10.1038/nrrheum.2013.7. Epub 2013 Feb 19. PMID 23419429
- [Background] Ghoreschi K, Jesson MI, Li X, Lee JL, Ghosh S, Alsup JW, Warner JD, Tanaka M, Steward-Tharp SM, Gadina M, Thomas CJ, Minnerly JC, Storer CE, LaBranche TP, Radi ZA, Dowty ME, Head RD, Meyer DM, Kishore N, O'Shea JJ. Modulation of innate and adaptive immune responses by tofacitinib (CP-690,550). J Immunol. 2011 Apr 1;186(7):4234-43. doi: 10.4049/jimmunol.1003668. Epub 2011 Mar 7. PMID 21383241
- [Derived] Hasni SA, Gupta S, Davis M, Poncio E, Temesgen-Oyelakin Y, Carlucci PM, Wang X, Naqi M, Playford MP, Goel RR, Li X, Biehl AJ, Ochoa-Navas I, Manna Z, Shi Y, Thomas D, Chen J, Biancotto A, Apps R, Cheung F, Kotliarov Y, Babyak AL, Zhou H, Shi R, Stagliano K, Tsai WL, Vian L, Gazaniga N, Giudice V, Lu S, Brooks SR, MacKay M, Gregersen P, Mehta NN, Remaley AT, Diamond B, O'Shea JJ, Gadina M, Kaplan MJ. Phase 1 double-blind randomized safety trial of the Janus kinase inhibitor tofacitinib in systemic lupus erythematosus. Nat Commun. 2021 Jun 7;12(1):3391. doi: 10.1038/s41467-021-23361-z. PMID 34099646
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-AR-0185.html